CLINICAL TRIAL: NCT03461484
Title: A French Post-market Observational/Non-interventional Study of the BioMatrix Flex™ and BioMatrix Neo Flex™ Drug Eluting Stents With 6-month DAPT
Brief Title: e-BioMatrix 6 Month DAPT France
Status: Completed | Type: Observational
Sponsor: Biosensors Europe SA (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: 13-EU-02
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Stenoses; Stable Angina; Ischemia; NSTEMI - Non-ST Segment Elevation MI; STEMI
MeSH Terms: conditions — Coronary Stenosis; Angina, Stable; Ischemia; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, multi-center observational study to be conducted in up to 30 French interventional cardiology centers. The purpose of this observational study is to capture, in French Centers, clinical data of the BioMatrix Flex™ and BioMatrix NeoFlex™ Drug Eluting Coronary Stents System (Biolimus A9, BA9™-) in normal practice, in patients treated with 6-month DAPT, and to compare the outcomes to those of previous e-biomatrix registries with longer DAPT durations. The patients will be followed up for 2 years for data collection.

ELIGIBILITY:
Inclusion Criteria:

* "Real world, all comer" patients

  1. Age ≥18 years;
  2. Patients that need a treatment with a BioMatrix Flex™ drug- eluting stent or a BioMatrix NeoFlex™drug-eluting stent;
  3. Presence of one or more coronary artery stenoses in a native coronary artery from 2.25 to 4.0 mm in diameter that can be covered with one or multiple stents;
  4. No limitation on the number of treated lesions, vessels, and lesion length, within the limits of social security reimbursements;
  5. Patient with DAPT indication after PCI.

Exclusion Criteria:

1. Inability to provide informed consent;
2. Patients needing additional stent NOT of the BioMatrix Flex™ or NeoFlex™ types;
3. Patients receiving next to the BioMatrix Flex™ or BioMatrix NeoFlex™ also other coronary vascular interventions, for example, balloon dilation;
4. Pregnant or planning to become pregnant patient;
5. DES and BMS implantation less than 6 months before screening;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "Real world, all comers" patient population: Patients with symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes, who qualify for percutaneous coronary interventions and can be treated with 6-month DAPT
Sampling Method: Non-Probability Sample
Enrollment: 2098 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) in the overall population, defined as composite of all-cause death, cerebrovascular accidents, non fatal myocardial infarction or clinically-driven target vessel revascularization at 6 months | 6 months
  Major adverse cardiac and cerebrovascular events (MACCE) in the overall population, defined as composite of all-cause death, cerebrovascular accidents, non fatal myocardial infarction or clinically-driven target vessel revascularization at 6 months

SECONDARY OUTCOMES:
Primary and secondary stent thrombosis | 6 months and 2 years
  Primary and secondary stent thrombosis (definite and probable according to ARC definitions) at 6 months and 2 years;
Major bleeding | 6 months and 2 years
  Major bleeding (BARC 3, 4 and 5 definitions) at 6 months and 2 years
Major adverse cardiac and cerebrovascular events (MACCEs) in the overall population | 2 years
  Major adverse cardiac and cerebrovascular events (MACCEs) in the overall population, defined as composite of all cause death, myocardial infarction (Q-wave and non-Q-wave), cerebrovascular accidents or clinically-driven target vessel revascularization at 2 years
Cardiac deaths at 6 months and and 2 years | 6 months and and 2 years
  Cardiac deaths at 6 months and and 2 years
Patient Oriented Composite Endpoint defined as any cause mortality, MI (Q-wave and non-Q-wave), or any revascularization at 6 months and 2 years | 6 months and 2 years
  Patient Oriented Composite Endpoint defined as any cause mortality, MI (Q-wave and non-Q-wave), or any revascularization at 6 months and 2 years
Death,MI and cerebrovascular accidents at 6 months and 2 years | 6 months and 2 years
  Death,MI and cerebrovascular accidents at 6 months and 2 years
Death, post-procedural MI and cerebrovascular accidents at 6 months and 2 years | 6 months and 2 years
  Death, post-procedural MI and cerebrovascular accidents at 6 months and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Spaulding, MD, Principal Investigator — Hôpital Européen Georges-Pompidou; Lanusz Lipiecki, MD, Principal Investigator — Clinique des Dômes

IPD SHARING:
Plan to Share IPD: No
Not planned